CLINICAL TRIAL: NCT05707624
Title: Randomized Controlled Study: The Effect of Distance Education Given With the Video Prepared for the Approach to the Febrile Child on the Knowledge, Attitudes and Behaviors of the Parents.
Brief Title: The Effect of Video Education to the Febrile Child on the Knowledge, Attitudes and Behaviors of the Parents.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Fatma Toksöz, Research Assistant, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 13895138840
Record Dates: First submitted 2022-12-26; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Fever; Child, Only; Approach-Approach Conflict; Parents
MeSH Terms: conditions — Fever

STUDY DESIGN:
Intervention Model Description: Simple random sampling method was used in the study. Parents who met the research inclusion criteria were assigned to the groups by drawing lots. In the lottery method, first of all, the control and intervention groups were written by the researcher on 1st paste and 80 g/m2 A4 papers of 4x4 cm size and the papers were placed in a bag that is invisible. Then, when the first parent who met the criteria for inclusion in the emergency room came, any nurse working in the service other than the researcher was asked to choose a paper from the bag (by blinding). If a control group is written on the paper, it is assigned to the parent control group, and if it is written as an intervention group, it is assigned to the parent intervention group. When the second parent who met the criteria for inclusion in the emergency department came, lots were not drawn, and the parent was assigned to the other group. The same procedure was repeated for all subsequent participants.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): During the process; Phone numbers were obtained and recorded at the first meeting with the parents. The link of the first two training videos was sent to the smartphones of the participants at the same time. Parents are explained how to access the videos from the link. Afterwards, other training videos, prepared once a week and as 2 videos, were sent to the parents' smartphones on a regular basis.
  After the procedure; Participants were contacted by phone 2 weeks after the last videos were watched. They were asked to fill out and send the questionnaire and scale online sent to their phones.
  Interventions: Other: video education
- Control group (Placebo Comparator): During the process; The phone number obtained from the parents was recorded and no other application was made other than the routine procedure of the clinic. Parents were not contacted in the following weeks.
  After the procedure; The control group was also reached via telephone 2 weeks after the video submission to the intervention group was completed. They were asked to fill out and send the questionnaire and scale online sent to their phones.
  Interventions: Other: the routine procedure

INTERVENTIONS:
Other: video education — In the study, there are 2 groups in total: the intervention group (n=50) which videos of approaching the febrile child was watched once a week and 2 videos, and the control group (n=49) which no other application is made except for the routine procedure of the hospital
  Arms: experimental
Other: the routine procedure — the routine procedure
  Arms: Control group

SUMMARY:
Aim: The study was carried out to evaluate the effect of distance education, which is given with a video prepared for the approach to the child with fever, on the knowledge, attitudes and behaviors of parents with children in the 0-5 age group.

Method: This is a randomized controlled intervention study. The research was carried out in Eskişehir City Hospital Pediatric Emergency Service, between 8th April 2022 and 10th June 2022. The study was completed with 99 parents with children aged 0-5 years old who consulted to the pediatric emergency service with the complaint of fever. In the study, there are 2 groups in total: the intervention group (n=50) which videos of approaching the febrile child was watched once a week and 2 videos, and the control group (n=49) which no other application is made except for the routine procedure of the hospital. "Descriptive Information Form" and "Parental Fever Management Scale" were used to collect data. Data collection tools were applied to the parents before and after the application. IBM SPSS Statistics 26 package program was used to evaluate the data. A statistically significant p<0.05 value was accepted.

DETAILED DESCRIPTION:
Introduction and Purpose:

Fever is a condition that occurs as a result of the deterioration of the balance between heat production and consumption in the body (Crisp et al., 2016). Fever is not a disease in itself, but one of the defense mechanisms of the body that arises due to diseases (Crisp et al., 2016; Karaca Çiftçi & Beklen, 2014). Fever complaints constitute the majority of pediatric emergency service applications (Esenay et al., 2007; Karakaş et al., 2020; Saz et al., 2009). Parents think that the fever will harm their children and they are afraid that they will have a seizure. The biggest factor underlying this fear is that parents do not have enough information about fever and fever management. Studies (Çöl Araz, 2013; Eliçık et al., 2012; Kılıç et al., 2016; Kılıçaslan et al., 2018) revealed that parents lack information on fever measurement, normal limits of fever, causes of fever, methods of reducing fever, and drug doses. shows that they need training on these issues.n addition, many parents may make wrong practices in order to reduce the fever of the child at home (Karaca Çiftçi & Beklen, 2014; Thota et al., 2018; Wilson et al., 2019). Nurses have the greatest responsibility in this regard. Because nurses have the opportunity to work with individuals in many environments such as schools, workplaces, hospitals, and they are the health professionals who can reach the society most easily. Nurses should identify the knowledge deficiencies of individuals in every environment they are in and try to eliminate them with education (Aydemir Geduk, 2018). However, it has been determined in the literature (Dinçer & Arslan, 2017; Sökün & Gözen, 2017) that nurses also need information about approaching children with fever. The lack of a common consensus in the approach to the child with fever may lead individuals to make wrong practices. For this purpose, it is important to follow the current and evidence-based literature on the approach to the child with fever (NICE, 2019; Toksöz & Açıkgöz, 2022). In addition, technology can be used to make education accessible to wider audiences and to be accessible at any time.In addition, making use of evidence-based research and guidelines can lead to the adoption of a common approach. This study was carried out to evaluate the effect of distance education, which is given with a video prepared for the approach to the child with fever, on the knowledge, attitudes and behaviors of parents who have children in the 0-5 age group, in line with current and evidence-based studies.

Method: This is a randomized controlled intervention study.

Dependent variables of the study: "Parental Fever Management Scale" score, parents' knowledge levels about fever and their knowledge, attitudes and behaviors about fever.

Independent variables of the research: "Educational Videos for Approaching Children with Fever", socio-demographic characteristics of parents.

his is a randomized controlled intervention study. The research was carried out in Eskişehir City Hospital Pediatric Emergency Service, between 8th April 2022 and 10th June 2022. The study was completed with 99 parents with children aged 0-5 years old who consulted to the pediatric emergency service with the complaint of fever. In the study, there are 2 groups in total: the intervention group (n=50) which videos of approaching the febrile child was watched once a week and 2 videos, and the control group (n=49) which no other application is made except for the routine procedure of the hospital. "Descriptive Information Form" and "Parental Fever Management Scale" were used to collect data. Data collection tools were applied to the parents before and after the application. IBM SPSS Statistics 26 package program was used to evaluate the data. A statistically significant p<0.05 value was accepted.

Sampling inclusion criteria:

The parent brought the child to the emergency room with a complaint of fever, The child is between 0-5 years old, Parent's consent to participate in the study, Parent's ability to read and write, Parent's ability to understand and speak Turkish, Parent has a smartphone to watch videos

Exclusion criteria:

If the parent has a disability that will prevent them from participating in the training (For example, having a hearing impairment, etc.) The age of the child is over 5 years old.

Data Collection Tools:

In data collection; Descriptive Information Form and Parental Fever Management Scale (Pfms-Tr) were used. In addition, the Global Quality Scoring System was used to evaluate the content of educational videos for children with fever, and the Journal of American Medical Association Benchmark Criteria was used to evaluate video resources.

Ethical Aspect of Research:

Before starting the research, T.C. Ethics committee approval (dated 17 June 2021 and numbered E-80558721-050.99-194226) was received from Eskişehir Osmangazi University Clinical Research Ethics Committee. In addition, institutional permission (dated 10.03.2022 and numbered E-11202945-605.01) was obtained from the Eskişehir Provincial Health Directorate for the hospital where the research would be conducted. In the study, verbal and written consent was obtained from the parents after informing them. Permission to use the scale was obtained from the owner of the scale who made the Turkish version of the Parental Fever Management Scale used in the study.

ELIGIBILITY:
Inclusion Criteria:

* The parent brought the child to the emergency room with a complaint of fever,
* The child is between 0-5 years old,
* Parent's consent to participate in the study,
* Parent's ability to read and write,
* Parent's ability to understand and speak Turkish,
* Parent has a smartphone to watch videos.

Exclusion Criteria:

* If the parent has a disability that will prevent them from participating in the training (For example, having a hearing impairment, etc.)
* The age of the child is over 5 years old.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
descriptive information form | 2 months
  This form measures participants knowledge, attitude and behaviours about fever in 0-5 ages children. After intervention, it is expected that; The intervention group which was given remote video training for fever, had a higher level of knowledge and positive attitudes and behaviours about fever than the control group, where the routine procedure of the hospital was applied.
Parent fever management scale | 2 months
  This scale measures patients fever management for their children. It shows that parents have more fever anxiety and perform more fever management when the scale scores are high.
  After intervention, it is expected that; The Parental Fever Management Scale scores of the intervention group given remote video training for fever were lower than the control group in which the routine procedure of the hospital was applied.

CONTACTS AND LOCATIONS:
Overall Officials: fatma Toksoz, Study Director — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Tepebasi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toksoz F, Acikgoz A. Randomized controlled study: The effect of video-based distance education for approaching children with fever on parents' knowledge levels and fever management. J Pediatr Nurs. 2024 May-Jun;76:e42-e49. doi: 10.1016/j.pedn.2024.01.017. Epub 2024 Jan 25. PMID 38278747